CLINICAL TRIAL: NCT06964035
Title: Influence of Original Native Aortic Valve Lesion (Stenosis or Steno-insufficiency vs. Insufficiency) on Post-implant Structural Bioprosthetic Degeneration After Aortic Valve Replacement
Acronym: DURABLE-AORTIC
Status: Enrolling by invitation | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Roberto Lorusso, Prof. MD PhD, Maastricht University Medical Center
Other Study IDs: METC 2023-0326
Record Dates: First submitted 2025-03-07; First posted 2025-05-09 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Aortic Bioprosthesis Degeneration
Keywords: aortic bioprosthesis; bioprosthesis degeneration
MeSH Terms: interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All patients undergoing elective aortic valve replacement for stenotic aortic valve replacement or a: All patients undergoing elective aortic valve replacement for stenotic aortic valve replacement or aortic valve regurgitation at our institution from 2012 to 2021 who met the inclusion criteria for the study (described in the dedicated session) will be enrolled in the study
  Interventions: Procedure: Aortic valve replacement

INTERVENTIONS:
Procedure: Aortic valve replacement — All operations were performed through median longitudinal sternotomy or mini-sternotomy.
  8 Intraoperative transesophageal echocardiography (TOE) was used in all patients. Arterial cannulation was central and venous cannulation was achieved with a common two-stage cannula in the right atrium. Left ventricle was vented through the right superior pulmonary vein. In minimally invasive procedures, venous cannulation was achieved percutaneously. Myocardial protection was achieved by administration of cold crystalloid or blood cardioplegia at the surgeon's discretion in an antegrade (indirect or selective) or retrograde fashion. The removal of the calcified cusps and the decalcification of the annulus was performed according to traditional techniques. All the prosthesis were be implanted with supranular technique and 2-0 U-shaped pledgeted sutures.

SUMMARY:
All patients undergoing elective aortic valve replacement for stenotic aortic valve replacement or aortic valve regurgitation at our institution from 2012 to 2021 who met the inclusion criteria for the study (described in the dedicated session) will be enrolled in the study. These patients will be contacted to provide information about the clinical status, NYHA functional class, possible rehospitalization, possible cardiovascular events and to perform a postoperative echocardiography if not performed in the previous year. Once consent is given, pre-, intra- and post-operative data will be collected in a dedicated, structured, database.

DETAILED DESCRIPTION:
All patients undergoing elective aortic valve replacement for stenotic aortic valve replacement or aortic valve regurgitation at our institution from 2012 to 2021 who met the inclusion criteria for the study (described in the dedicated session) will be enrolled in the study. These patients will be contacted to provide information about the clinical status, NYHA functional class, possible rehospitalization, possible cardiovascular events and to perform a postoperative echocardiography if not performed in the previous year. Once consent is given, pre-, intra- and post-operative data will be collected in a dedicated, structured, database.

ELIGIBILITY:
Inclusion Criteria:

* - Age ≥ 18 years; 9
* Patients who underwent isolated aortic and mitral valve replacement for stenosis or regurgitation
* Signed informed consent, inclusive of release of medical information.

Exclusion Criteria:

* - Aortic and mitral valve replacement associated with surgery of ascending aorta/aortic root;
* Aortic and mitral valve replacement associated with other cardiac valve surgery (apart from arrythmia-related ablation or procedures);
* Previous cardiac surgery of any kind;
* Surgery for acute endocarditis
* Surgery for Type A aortic dissection
* Participation in another clinical trial that could interfere with the endpoints of this study.
* Pregnant or breastfeeding at time of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing elective aortic valve replacement for stenotic aortic valve replacement or aortic valve regurgitation at our institution from 2012 to 2021 who met the inclusion criteria for the study (described in the dedicated session) will be enrolled in the study. These patients will be contacted to provide information about the clinical status, NYHA functional class, possible rehospitalization, possible cardiovascular events and to perform a postoperative echocardiography if not performed in the previous year. Once consent is given, pre-, intra- and post-operative data will be collected in a dedicated, structured, database.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Prosthetic valve deterioration and degenration | 10-15 years
  Echocardiographic analisys with multiparametric datas will be used. From quantitative to qualitative.

SECONDARY OUTCOMES:
Survival | 15 years
  Longitudinal analysis will be used to establish the surival rate at long term.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht UMC+ METC, Maastricht, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided